CLINICAL TRIAL: NCT03253627
Title: Mindfulness-Based Stress Reduction To Improve Cognitive Function for Postmenopausal Women With Breast Cancer
Brief Title: MBSR During AI Therapy for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: s17-00995; 4R00NR015473-03 (NIH)
Record Dates: First submitted 2017-08-08; First posted 2017-08-18 (Actual); Results first posted 2022-05-19 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer; Cognitive Symptom
MeSH Terms: conditions — Breast Neoplasms; Neurobehavioral Manifestations | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: A pilot, single-center randomized controlled trial of the preliminary efficacy of an eight-week, group-based Mindfulness-Based Stress Reduction intervention versus Health Enhancement Program active control (i.e., two groups, parallel design) to improve neural markers of changes in cognitive function in postmenopausal women receiving aromatase inhibitor therapy for breast cancer. Participants will be stratified in a permuted block design by receipt of chemotherapy (i.e., two strata). Data will be collected at up to three time points using a repeated measures design (i.e., pre-intervention, post-intervention, approximately three months after the intervention). The study groups will meet at NYU for MBSR or HEP. Neuropsychological, self-report, and biospecimen data collection will be conducted at the Bluestone Center. Neuroimaging data will be collected at the NYU Center for Brain Imaging.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will complete the baseline assessment and be randomly assigned to study group in a permuted block design stratified by receipt of chemotherapy (i.e., two strata). It will not be possible to blind study participants or interventionists to group assignment. To reduce bias, research staff who conduct assessments, including the PI, will be blinded to group assignment (i.e., single blind). Participants will be reminded not to reveal their group assignment to study staff conducting assessments. The study biostatistician will have no direct contact with study participants and will not be blinded to group assignment. The biostatistician will produce and maintain the randomization codes for the permuted blocks. Randomization may only be unmasked by the biostatistician at the completion of data collection, or for reporting of serious adverse events or unanticipated problems for which it will be essential to provide information to the PI on group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR (Experimental): Mindfulness-Based Stress Reduction
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Health Enhancement Program (Active Comparator): Health Enhancement Program
  Interventions: Behavioral: Health Enhancement Program

INTERVENTIONS:
Behavioral: Health Enhancement Program — The HEP control, which was developed to serve as an active control to MBSR, will receive manualized health education from experts in physical activity, functional movement, music therapy, and nutrition-without mindfulness instruction-using similar modalities to MBSR training for a matched schedule.
  Other Names: HEP
  Arms: Health Enhancement Program
Behavioral: Mindfulness-Based Stress Reduction — The MBSR group will receive training from a certified instructor during a group-based, 2.5-hour manualized educational activity weekly for eight weeks. Activities include body scans, gentle stretching, yoga, and mindful awareness. Participants will be asked to complete daily 45-minute, audio-guided mindfulness activities and a one-day weekend retreat to reinforce learning.
  Other Names: MBSR
  Arms: MBSR

SUMMARY:
This study will use non-invasive neuroimaging (i.e., MRI) to examine whether Mindfulness-Based Stress Reduction (MBSR) improves neural markers of cognitive function for postmenopausal women taking aromatase inhibitor (AI) therapy for breast cancer. The pilot randomized controlled trial will obtain preliminary efficacy of MBSR versus Health Enhancement Program (HEP) active control to improve neural markers of cognitive function. The final sample will include 32 postmenopausal women with breast cancer. MBSR and HEP groups will meet for a matched schedule of 8 weekly 2.5-hour sessions and a one-day weekend retreat. Specimen and data collection will be done at three time points: pre-randomization (i.e., within three weeks before beginning the intervention), within three weeks after completion of the intervention, and approximately three months (+/- three weeks) post intervention. Change scores for neuroimaging parameter estimates will be correlated with change scores for measures of cognitive function and affect. Differential expression of genes will be correlated with neuroimaging parameter estimates.

DETAILED DESCRIPTION:
Adjuvant aromatase inhibitor (AI) therapy improves disease-free and overall survival for postmenopausal women after surgery for hormone receptor-positive breast cancer. Among symptoms associated with AI therapy are changes in cognitive function. Up to 25% of postmenopausal women with breast cancer report that they experience changes in cognitive function during AI therapy. Studies using neuropsychological tests found subtle deteriorations in verbal and visual learning and memory-as well as concentration, working memory, and executive function-for as many as a third of these patients. Changes in cognitive function may be associated with changes in affect (e.g., worry, depressive symptoms). Neural markers of cognitive changes, including changes in brain function and structure, may underlie changes in cognitive function.

The investigators' recent preliminary neuroimaging work to describe neural markers of cognitive changes suggests that postmenopausal women with breast cancer have inefficient cognitive-emotion processing before AI therapy, as evidenced by greater neural activity in the hippocampus (working memory) and amygdala (emotion processing) during task performance compared to controls. During AI therapy, patients show differential activation compared to controls in the dorsolateral prefrontal cortex (executive function and working memory), medial prefrontal cortices (cortical control of amygdala responses), and hippocampus.

Stress responses could partially explain relationships between AI therapy and neural markers of cognitive changes. The Mindfulness Stress-Buffering Account suggests that interventions such as Mindfulness-Based Stress Reduction (MBSR) may improve stress responses by attenuating negative appraisals of stress and reducing reactivity to stressful situations. For example, mindfulness meditation improved psychological stress responses in women with breast cancer. It improved some measures of cognitive function. Mindfulness practices reduced physiological markers of stress responses, including inflammatory markers in women with breast cancer and in stressed community adults, as well as cortisol reactivity for breast cancer survivors and during chemotherapy for colorectal cancer. Although similar neural deficits as were found in the investigators' preliminary work have been shown to improve in stressed adult populations using MBSR, it is not known whether the intervention improves neural deficits in women taking AI therapy (estrogen, production of which is blocked by AI therapy, is neuroprotective and promotes neural plasticity). Genetic variability was previously found to moderate the effect of MBSR on self-reported cognitive function. Therefore, it is possible that inter-individual variability in the expression of genes involved in stress responses could moderate relationships between AI therapy and neural markers of cognitive changes during MBSR. Taken together, MBSR may improve neural markers of cognitive changes shown in preliminary work to be deficient in postmenopausal women before and during AI therapy for breast cancer by targeting stress responses. Changes in these neural markers may correspond to improved self-report and neuropsychological measures of cognitive function.

Hypothesis: Stress reduction, moderated by gene expression, blunts the impact of AI therapy on neural markers of cognitive function, thereby improving cognitive function and affect in women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. <80 years of age by date of baseline assessment visit
3. Able to speak and read English
4. Post-menopausal (defined as [A] amenorrhea persisting for an entire year, [B] oophorectomy or ovarian suppression/ablation, or [C] hysterectomy and age >51 years)
5. Diagnosed with DCIS (stage 0) or stage I, II, or III breast cancer
6. Post lumpectomy or mastectomy and any re-excisions
7. Post neoadjuvant or adjuvant chemotherapy, if prescribed
8. Taking aromatase inhibitor (AI) therapy OR AI therapy scheduled to begin before planned post-intervention assessment visit

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer
2. Diagnosis of a major psychiatric disorder (e.g., bipolar I disorder, schizophrenia, schizoaffective disorder)
3. Suicide attempt within the last 10 years
4. Hospitalization or residential treatment for psychiatric illness, eating disorder, or substance abuse within the last 2 years
5. History of neurological disease (e.g., Parkinson's disease, dementia)
6. History of head trauma
7. Claustrophobia
8. Unable to lie on the back
9. Ever been told not to get an MRI
10. MRI-incompatible metal implant*

    * If a potential participant reports implanted metal objects, which might be affected by MRI magnets, the study personnel and MRI technologist will screen over the phone or in person to determine whether the potential participant would be safe during the MRI scan. A current list of implants compatible with MRI will be consulted (http://www.mrisafety.com/TMDL_list.php).

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Merriman, PhD, RN, Principal Investigator — New York University Meyers College of Nursing
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Even though the R00 study is not anticipated to reach the threshold for required genomic data sharing, the study will have in place plans for sharing de-identified data for secondary analyses with qualified investigators. The consent language for the R00 study will be worded for possible broad data sharing.
Time Frame: The timeline for submission to an NIH-designated data repository will allow first for publication of findings related to the aims of the R00 study, as well as submission of findings as preliminary data for anticipated grant application(s).
Access Criteria: The investigators plan to submit genomic data and relevant phenotypic data (e.g., clinical characteristics of the sample) generated in the R00 study to an NIH-designated data repository in a timely manner. The submission process will likely include registration in the database of Genotypes and Phenotypes (dbGaP) and submission to Gene Expression Omnibus (GEO) for controlled access to the data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: NYU was activated as a site in September 2017. Recruitment and screening began in January 2018. Enrollment started in April 2018 and ended in October 2019. Bellevue Hospital site approval was received in July 2019. Enrollment began then in its affiliated clinics and ended in October 2019.
Period: Overall Study
Arm/Group | MBSR | Health Enhancement Program
Started | 12 | 11
Post-intervention | 11 | 9
Completed | 10 | 7
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Inability to complete MRI | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MBSR | Health Enhancement Program | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (4.85) | 55.6 (10.51) | 61 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 10 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Functional Neural Activation Parameter Estimate
Description: global maximum cluster-level neural activation during task-based functional magnetic resonance imaging for MBSR group compared to Health Enhancement Program group in a whole-brain analysis; paradigm: Emotional Faces N-Back; conditions: happy face distractors minus no face distractors; value has no minimum or maximum; value has no reference ranges; higher values indicate more neural activation
Time Frame: baseline, 3 months
Population: participants with usable neuroimaging data after quality control
Measure: Mean (Standard Deviation); unit: beta weights
Arm/Group | MBSR | Health Enhancement Program
Number analyzed (Participants) | 10 | 8
beta weights
  baseline | -1.2 (2.27) | -1.8 (2.28)
  3 months | -0.8 (1.95) | -0.7 (2.27)
Statistical Analysis 1: Comparison: MBSR vs Health Enhancement Program; baseline; Test type: Superiority; p = 0.460, t-test, 2 sided
Statistical Analysis 2: Comparison: MBSR vs Health Enhancement Program; 3 months; Test type: Superiority; p = 0.896, t-test, 2 sided

2. Other Pre Specified Outcome: List Sorting Working Memory Test
Description: from National Institutes of Health (NIH) Toolbox; Age 7+ v2.1; measures working memory; T-score range 23-77; 50 indicates the population mean with a standard deviation of 10; higher scores indicate better working memory performance; scores below 40 suggest cognitive impairment
Time Frame: baseline, 6 months
Population: differences in sample size due to attrition
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | MBSR | Health Enhancement Program
Number analyzed (Participants) | 12 | 11
T-score
  baseline | 48.7 (6.05) | 51.5 (8.57)
  6 months: number analyzed (Participants) | 10 | 7
  6 months | 50.5 (8.57) | 56.3 (10.75)
Statistical Analysis 1: Comparison: MBSR vs Health Enhancement Program; baseline; Test type: Superiority; p = 0.374, t-test, 2 sided
Statistical Analysis 2: Comparison: MBSR vs Health Enhancement Program; 6 months; Test type: Superiority; p = 0.236, t-test, 2 sided

3. Other Pre Specified Outcome: Flanker Inhibitory Control and Attention Test
Description: from National Institutes of Health (NIH) Toolbox; Age 12+ v2.1; measures attention; T-score range 23-77; 50 indicates the population mean with a standard deviation of 10; higher scores indicate better attention performance; scores below 40 suggest cognitive impairment
Time Frame: baseline, 6 months
Population: Differences in sample size due to attrition
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | MBSR | Health Enhancement Program
Number analyzed (Participants) | 12 | 11
T-score
  baseline | 46.5 (8.17) | 41.9 (7.64)
  6 months: number analyzed (Participants) | 10 | 7
  6 months | 43.3 (3.83) | 42.4 (11.27)
Statistical Analysis 1: Comparison: MBSR vs Health Enhancement Program; baseline; Test type: Superiority; p = 0.180, t-test, 2 sided
Statistical Analysis 2: Comparison: MBSR vs Health Enhancement Program; 6 months; Test type: Superiority; p = 0.822, t-test, 2 sided

4. Other Pre Specified Outcome: Cognitive Function
Description: From the Quality of Life in Neurological Disorders (Neuro-QoL) Bank; v2.0; patient-reported outcome; measures executive function and general cognitive concerns; T-score range 17.3-64.2; 50 indicates the population mean with a standard deviation of 10; higher scores indicate better self-reported cognitive function; scores 41-45 suggest mild cognitive impairment, 31-40 suggest moderate cognitive impairment, and 30 or below suggest severe cognitive impairment
Time Frame: baseline, 3 months, 6 months
Population: Differences in sample size due to attrition
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | MBSR | Health Enhancement Program
Number analyzed (Participants) | 12 | 11
T-score
  baseline | 47.0 (6.49) | 45.9 (8.20)
  3 months: number analyzed (Participants) | 11 | 9
  3 months | 45.4 (5.12) | 46.0 (8.93)
  6 months: number analyzed (Participants) | 10 | 7
  6 months | 47.4 (6.37) | 46.4 (7.57)
Statistical Analysis 1: Comparison: MBSR vs Health Enhancement Program; baseline; Test type: Superiority; p = .715, t-test, 2 sided
Statistical Analysis 2: Comparison: MBSR vs Health Enhancement Program; 3 months; Test type: Superiority; p = 0.861, t-test, 2 sided
Statistical Analysis 3: Comparison: MBSR vs Health Enhancement Program; 6 months; Test type: Superiority; p = .790, t-test, 2 sided

5. Other Pre Specified Outcome: Anxiety
Description: From the Quality of Life in Neurological Disorders (Neuro-QoL) Bank; v1.0; patient reported outcome; T-score range 36.4-76.8; 50 indicates the population mean with a standard deviation of 10; higher scores indicate worse self-reported anxiety; scores 55-59 suggest mild anxiety, 60-69 suggest moderate anxiety, and 70 or above suggest severe anxiety
Time Frame: baseline, 3 months, 6 months
Population: Differences in sample size due to attrition
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | MBSR | Health Enhancement Program
Number analyzed (Participants) | 12 | 11
T-score
  baseline | 51.3 (5.40) | 53.1 (5.96)
  3 months: number analyzed (Participants) | 11 | 9
  3 months | 48.8 (6.91) | 53.9 (12.28)
  6 months: number analyzed (Participants) | 10 | 7
  6 months | 46.7 (7.56) | 50.3 (12.66)
Statistical Analysis 1: Comparison: MBSR vs Health Enhancement Program; baseline; Test type: Superiority; p = 0.452, t-test, 2 sided
Statistical Analysis 2: Comparison: MBSR vs Health Enhancement Program; 3 months; Test type: Superiority; p = 0.253, t-test, 2 sided
Statistical Analysis 3: Comparison: MBSR vs Health Enhancement Program; 6 months; Test type: Superiority; p = 0.469, t-test, 2 sided

6. Other Pre Specified Outcome: Depression
Description: From the Quality of Life in Neurological Disorders (Neuro-QoL) Bank; v1.0; patient-reported outcome; measures depressive symptoms; T-score range 36.9-75.0; 50 indicates the population mean with a standard deviation of 10; higher scores indicate worse depressive symptoms; scores 55-59 suggest mild depressive symptoms, 60-69 suggest moderate depressive symptoms, and 70 or above suggest severe depressive symptoms
Time Frame: baseline, 3 months, 6 months
Population: Differences in sample size due to attrition
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | MBSR | Health Enhancement Program
Number analyzed (Participants) | 12 | 11
T-score
  baseline | 46.3 (6.31) | 45.3 (3.24)
  3 months: number analyzed (Participants) | 11 | 9
  3 months | 46.0 (6.78) | 49.7 (10.41)
  6 months: number analyzed (Participants) | 10 | 7
  6 months | 44.9 (7.24) | 48.4 (8.91)
Statistical Analysis 1: Comparison: MBSR vs Health Enhancement Program; baseline; Test type: Superiority; p = 0.628, t-test, 2 sided
Statistical Analysis 2: Comparison: MBSR vs Health Enhancement Program; 3 months; Test type: Superiority; p = 0.345, t-test, 2 sided
Statistical Analysis 3: Comparison: MBSR vs Health Enhancement Program; 6 months; Test type: Superiority; p = 0.384, t-test, 2 sided

7. Other Pre Specified Outcome: Gene Expression
Description: AMIGO1 gene expression in raw gene counts for MBSR group compared to Health Enhancement Program group in a whole transcriptome analysis using ribonucleic acid sequencing (RNA-Seq); minimum 0, no maximum; value has no reference ranges; higher values indicate more gene expression
Time Frame: baseline, 3 months, 6 months
Population: participants with usable gene expression data after quality control
Measure: Mean (Standard Deviation); unit: raw gene counts
Arm/Group | MBSR | Health Enhancement Program
Number analyzed (Participants) | 9 | 9
raw gene counts
  baseline | 106.1 (74.98) | 137.3 (77.40)
  3 months: number analyzed (Participants) | 8 | 9
  3 months | 196.0 (210.74) | 176.3 (114.57)
  6 months: number analyzed (Participants) | 9 | 7
  6 months | 114.4 (81.11) | 218.3 (86.28)
Statistical Analysis 1: Comparison: MBSR vs Health Enhancement Program; baseline; Test type: Superiority; p = .398, t-test, 2 sided
Statistical Analysis 2: Comparison: MBSR vs Health Enhancement Program; 3 months; Test type: Superiority; p = 0.811, t-test, 2 sided
Statistical Analysis 3: Comparison: MBSR vs Health Enhancement Program; 6 months; Test type: Superiority; p = 0.027, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: For each participant, adverse event data were collected from the date of enrollment through the final assessment (i.e., approximately 6 months after enrollment).
Description: questionnaire at each follow-up assessment (i.e., post intervention, 3 months post intervention)
Arm/Group | MBSR | Health Enhancement Program
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

LIMITATIONS AND CAVEATS:
The sample was less than the anticipated final sample size of 32; it included fewer minority participants than planned. The advent of the COVID-19 pandemic prohibited further recruitment and conduct of this study, which had unavoidable in-person activities (e.g., neuroimaging).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT03253627/Prot_001.pdf
  • Statistical Analysis Plan (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT03253627/SAP_002.pdf
  • Informed Consent Form (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT03253627/ICF_000.pdf